CLINICAL TRIAL: NCT04380779
Title: Prevalence of Severe Bleeding in COVID-19 Patients Treated With Higher Than Recommended Thromboprophylaxis Doses (BLEEDING Study)
Brief Title: Prevalence of Severe Bleeding in COVID-19 Patients Treated With Higher Than Recommended Thromboprophylaxis Doses
Acronym: BLEEDING
Status: Completed | Type: Observational
Sponsor: Manuel Monreal (Other)
Responsible Party: Sponsor-Investigator, Manuel Monreal, Professor of Internal Medicine, Foundation for the study of VTE diseases. (FUENTE)
Organization: Foundation for the study of VTE diseases. (FUENTE) (Other)
Other Study IDs: BLEEDING042020
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objectives are:

* To establish the prevalence of major bleeding in patients treated with higher than recommended thromboprophylaxis doses.
* To identify variables associated to higher risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with COVID-19 treated with higher than recommended thromboprophylaxis doses.
* Admission to hospital.

Exclusion Criteria:

* Patients treated with ECMO (Extracorporeal membrane oxygenation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients infected with COVID-19 treated with higher than recommended thromboprophylaxis doses and admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 2430 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Bleeding events and complications | 30 days
  Study endpoints are clinically recognized (and objectively confirmed) major and minor bleeding complications, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Monreal, Study Chair — Germans Trias i Pujol Hospital
Locations (1):
- Manuel Monreal, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided